CLINICAL TRIAL: NCT02846038
Title: Understanding Communication in Healthcare to Achieve Trust (U-CHAT): A Prospective Longitudinal Investigation of Communication Between Pediatric Oncologists, Children/Adolescents With High-Risk Cancer, and Their Families at the Stressful Time-Points of Disease
Brief Title: Understanding Communication in Healthcare to Achieve Trust (U-CHAT)
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: U-CHAT; NCI-2021-10301 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Brain Tumors; Solid Tumor
Keywords: Pediatric cancer; Childhood cancer; High-risk disease; Prognosis; Communication; Bad news; Pediatric oncologist; Parent; Relapse; Progression
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Communication; Recurrence; Disease Progression

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient: Patients at St. Jude Children's Research Hospital who meet the eligibility criteria and consent to participate.
- Primary oncologist: Primary pediatric oncologists who meet the eligibility criteria and consent to participate.
- Parents of patient: Parents of the enrolled patient who meet eligibility criteria and consent to participate.

SUMMARY:
Honest, clear, and empathetic communication between pediatric oncologists (POs) and parents of children with cancer (POCCs) is imperative to facilitating therapeutic alliance and ensuring that medical management aligns with the families' goals of care. Communication is particularly important during conversations about disease reevaluation, which often necessitate parental decision-making in the context of emotional distress. POs employ a spectrum of communication styles and strategies during challenging conversations, and there is no consensus regarding linguistic or thematic metrics for high quality communication of upsetting information. In order to better understand how POs communicate difficult information to POCCs, the investigators propose a pilot study designed to accomplish the following primary aim:

Primary Objective:

* To identify recurrent verbal and nonverbal (e.g. the use of pauses/silence) communication techniques employed by POs in the delivery of difficult prognostic information to POCCs through content analysis of audio-recorded conversations between POs and parents of children with high risk cancer at the time of disease reevaluation.

The study expects to enroll up to: 80 patient participants, 80 parents, and 15 primary pediatric oncologists (total = 175).

Non-primary oncologist members of the clinical care team, extended family members, or friends of the family may also participate, if they choose to do so.

DETAILED DESCRIPTION:
Data collection will occur at each disease reevaluation, during which time the conversation will be audio-recorded and data will be abstracted from the medical record. Additionally, 2 surveys will be completed at specific time points by both the oncologist and the parent. Lastly, interviews will be offered to both the oncologist and the parent/patient following any audio-recorded conversation in which difficult news was discussed.

Disease reevaluation will be defined as any of the following interventions performed for the purposes of assessing disease status:

* Diagnostic imaging
* Lumbar puncture with cerebrospinal fluid analysis
* Bone marrow aspiration and/or biopsy
* Surgical biopsy or resection

The first time point for data collection with be at the time of the patient's first meeting with their oncologist to discuss the results of disease reevaluation. This discussion will be audio-recorded. The parent will be asked to complete a survey within 7 days. Those receiving difficult news will have the opportunity to participate in a brief interview with a study team member regarding their experience. Patients who are at least 12 years old will also have this opportunity, separate from their parents, if desired by the patient and approved by the parent. Interviews may be in person or by phone and have no set length.

The next time point for data collection will coincide with any time the patient/parents meet with their oncologist to discuss results of a disease reevaluation. Each conversation will be audio-recorded. If difficult news is delivered during the discussion, the parent and oncologist will be asked to complete a second survey for first bad news conversation, following the baseline recording. Parent, patient, and oncologist will be asked to participate in an interview for all bad news conversation.

Patient-parent dyads will be followed for a total of 24 months from the time of enrollment on study (defined as the date of first audio recording rather than date of actual consent), in the context of patients who do not experience disease relapse, progression, or refractory disease. Dyads in which patients experience disease relapse, progression, or refractory disease will be followed for a total of 24 months from the time of first disease relapse or progression while on study.

All data analyzed from audio-recordings will be permanently erased from recorders following completion of data analysis. Participants may request to discontinue to the study at any time.

For previously enrolled patients, (enrolled prior to revision 3.1), a retrospective chart review will be done to collect additional clinical data.

ELIGIBILITY:
Inclusion Criteria - Primary Oncologist:

* Primary oncologist is an attending physician (age 18+) who provides medical care to patients in the outpatient Solid Tumor or Neuro-Oncology clinics at St. Jude Children's Research Hospital.
* Primary hematology-oncology fellows (age 18+) who follow patients along with the primary oncologist will be eligible to participate in audio-recorded disease reevaluation conversations (and fellow contributions will be distinguished from primary oncologist contributions); however, they will not be eligible to complete post-conversation surveys nor semi-structured interviews.

Inclusion Criteria - Parents of Children with Cancer:

* Caregiver is 18 years of age or older.
* Caregiver is related to the patient in one of the following ways: biological parent, stepparent, or primary legal guardian.
* If more than 1 set of parents are involved, the caregiver with legal decision-making responsibilities will be eligible for participation.
* Caregiver is comfortable speaking and reading English.

Inclusion Criteria - Patients:

* Patient's primary oncologist is enrolled in this study.
* Patient (age ≤30 years) has been diagnosed with either a solid tumor and/or a brain tumor.
* Patient's primary pediatric oncologist documents or reports his/her impression that patient's likelihood of cure is 50% or less.
* Patient is projected to have ≥ 2 future time points of disease reevaluations, as documented in the electronic medical record (EMR) and/or confirmed by the patient's primary oncologist.
* Patient is being treated for one of the above high-risk diseases with <3 months until end-of-therapy disease evaluation, OR
* Patient's disease has relapsed, progressed, or not responded to therapy, as documented in the EMR and/or confirmed by the child's pediatric oncologist OR
* Patient is being treated for a uniformly fatal disease, such as diffuse intrinsic pontine glioma, or a disease in which the primary oncologist believes that the patient will almost certainly die, such as glioblastoma multiforme.

Inclusion Criteria - Non-Primary Oncologist Care Team Members, Patient's Extended Family Member, or Friend of the Family:

* Patient's primary oncologist is enrolled on the study.
* Patient's caregiver is enrolled on the study.
* Patient's caregiver has given verbal permission for non-primary oncologist clinical members of the patient's care team, the extended family member, or friend of the family to be present during the conversation between the patient's primary oncologist and the patient's caregiver.
* any non-primary oncologist members of the patient's clinical care team, the extended family members, or friends of the family (all age 18+ years) have all given verbal consent to be audio-recorded prior to the beginning of the conversation, in case they speak during the conversation between patient's primary oncologist and the patient's caregiver.

Exclusion Criteria:

* Implicitly stated in above inclusion criteria.
* Inability or unwillingness of potential research participant or legal guardian/representative to give informed consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from patients receiving care in the Solid Tumor or Neuro-Oncology clinics at St. Jude Children's Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Number of communication styles employed | From first patient visit for disease reevaluation through up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Erica Kaye, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols